CLINICAL TRIAL: NCT00222534
Title: Acetazolamide for Respiratory Failure in Combination With Metabolic Alkalosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oslo School of Pharmacy (Other)
Responsible Party: Principal Investigator, Torgeir Bruun Wyller, Professor, University of Oslo School of Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AREMA
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Respiratory Insufficiency; Alkalosis
Keywords: Respiratory Insufficiency; Alkalosis
MeSH Terms: conditions — Respiratory Insufficiency; Alkalosis | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Acetazolamide (Experimental): Acetazolamide 250 mg Three times a day for five days
  Interventions: Drug: Acetazolamide
- Placebo (Placebo Comparator): Placebo, one tablet Three times a day for five days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetazolamide
  Arms: Acetazolamide
Drug: Placebo
  Arms: Placebo

SUMMARY:
Respiratory failure is a common consequence of chronic obstructive pulmonary disease (COPD). A concurrent metabolic alkalosis may worsen the respiratory failure, as a higher pH in blood (and thus in cerebrospinal fluid) results in a weaker respiratory drive. Use of diuretics is the most common cause of metabolic alkalosis.

When a patient with an acute exacerbation of a respiratory failure is also alkalotic, there are (at least theoretical) reasons to lower the pH in order to increase the respiratory drive. Among other alternatives, the drug acetazolamide can be used for this purpose.

In some hospitals there is a tradition for the use of acetazolamide on this indication, but any evidence for the effect of such a treatment is rather weak.

Thus, the aim of this trial is to evaluate the effect of acetazolamide as an adjuvant treatment for hospitalized patients with acute exacerbation of respiratory failure in combination with metabolic alkalosis.

ELIGIBILITY:
Inclusion Criteria:

* Arterial pO2 8 kPa or lower, and arterial pCO2 7 kPa or higher.
* Base Excess 8 mmmol/l or higher.
* Written informed consent

Exclusion Criteria:

* Acetazolamide treatment regarded as obviously indicated or obviously contraindicated
* Already using acetazolamide
* Moribund patient
* Unable to give fully informed consent
* Allergy towards the tablet content or unable to swallow the tablets
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2002-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Partial pressure of oxygen in arterial blood on the 5th day of treatment (without extra oxygen)
Change in partial pressure of oxygen from start of treatment to the fifth day of treatment

SECONDARY OUTCOMES:
Partial pressure of carbon dioxide in arterial blood on the 5th day of treatment.
Change in partial pressure of carbon dioxide from start of treatment to the fifth day of treatment
Intrahospital deaths
Use of mechanical ventilation
Length of stay
Side effects

CONTACTS AND LOCATIONS:
Overall Officials: Torgeir B Wyller, MD, PhD, Principal Investigator — Department of Geriatric Medicine, Ullevaal University Hospital, Oslo, Norway
Locations (5):
- Norway (5):
  - Department of Respiratory Medicine, Haukeland University Hospital, Bergen
  - Department of Internal Medicine, Sorlandet Sykehus Kristiansand, Kristiansand
  - Department of Internal Medicine, Aker University Hospital, Oslo
  - Ullevaal University Hospital, Dept. of Respiratory Medicine, Oslo
  - Department of Internal Medicine, St.Olav's Hospital, Trondheim

REFERENCES:
- [Result] Gulsvik R, Skjorten I, Undhjem K, Holo L, Frostad A, Saure EW, Lejlic V, Humerfelt S, Hansen G, Bruun Wyller T. Acetazolamide improves oxygenation in patients with respiratory failure and metabolic alkalosis. Clin Respir J. 2013 Oct;7(4):390-6. doi: 10.1111/crj.12025. Epub 2013 Jul 4. PMID 23578004